CLINICAL TRIAL: NCT02624050
Title: Comparison of Methohexital With Propofol for Anesthetic Induction in Patients Treated With an Antagonist of the Renin-Angiotensin System.
Brief Title: Methohexital v Propofol as General Anesthetic in Patients on ACEIs or ARBs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Anthony Bonavia, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003830
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hypotension; Anesthesia
Keywords: ACEI; ARB; Hypotension; General Anesthesia; Methohexital; Propofol
MeSH Terms: conditions — Hypotension | interventions — Methohexital; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methohexital (Active Comparator): Methohexital will be administered intravenously as a general anesthetic at a dosage of 1.5mg per kg of patient body weight.
  Interventions: Drug: Methohexital
- Propofol (Active Comparator): Propofol will be administered intravenously as a general anesthetic at a dosage of 2.5mg per kg of patient body weight.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Methohexital — Both drugs of interest are standard of care for use as general anesthetics. The purpose of the study is the determine the susceptibility of both drugs to inducing a hypotensive event.
  Other Names: Brevital
  Arms: Methohexital
Drug: Propofol — Both drugs of interest are standard of care for use as general anesthetics. The purpose of the study is the determine the susceptibility of both drugs to inducing a hypotensive event.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
Patient undergoing general anesthesia in elective surgery will be assigned to receive either methohexital or propofol general anesthesia. Hypotensive events during the first 15 minutes of induction will be compared between the groups to ascertain which drug is less likely to cause a hypotensive event.

DETAILED DESCRIPTION:
Patients taking angiotensin converting-enzyme inhibitors (ACEIs) or angiotensin receptor blockers (ARBs) are susceptible to hypotensive events during general anesthesia. The purpose of this study is to determine if the use of either methohexital or propofol general anesthesias is more likely to result in hypotensive events in these patients during their induction. Hemodynamic metrics like blood pressure, mean arterial pressure, and heart rate will be monitored during the induction process, under both drugs, for use as the main metrics, as well as the need for vasopressors in response to patient hypotension.

ELIGIBILITY:
Inclusion Criteria:

* treated for at least 6 weeks with ACEIs or ARB
* undergoing elective surgery under general endotracheal anesthesia
* ASA Physical Class I or II

Exclusion Criteria:

* BMI >45kg/m^2
* taking both ACEI and ARB
* history of difficult intubation in the past
* require rapid sequence induction and intubation
* uncontrolled baseline blood pressure (SBP>180mmHg or DBP >110 mmHg) at anesthesia preoperative clinic visit
* contraindication to the use of propofol or methohexital
* significant coronary artery disease
* history of systolic heart failure
* history of renal failure (creatine level >2 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bonavia, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Ctr, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertrand M, Godet G, Meersschaert K, Brun L, Salcedo E, Coriat P. Should the angiotensin II antagonists be discontinued before surgery? Anesth Analg. 2001 Jan;92(1):26-30. doi: 10.1097/00000539-200101000-00006. PMID 11133595
- [Background] Carter JA, Clarke TN, Prys-Roberts C, Spelina KR. Restoration of baroreflex control of heart rate during recovery from anaesthesia. Br J Anaesth. 1986 Apr;58(4):415-21. doi: 10.1093/bja/58.4.415. PMID 3954922
- [Background] Cullen PM, Turtle M, Prys-Roberts C, Way WL, Dye J. Effect of propofol anesthesia on baroreflex activity in humans. Anesth Analg. 1987 Nov;66(11):1115-20. PMID 3499095
- [Background] Ebert TJ, Muzi M, Berens R, Goff D, Kampine JP. Sympathetic responses to induction of anesthesia in humans with propofol or etomidate. Anesthesiology. 1992 May;76(5):725-33. doi: 10.1097/00000542-199205000-00010. PMID 1575340
- [Background] Eyraud D, Brabant S, Nathalie D, Fleron MH, Gilles G, Bertrand M, Coriat P. Treatment of intraoperative refractory hypotension with terlipressin in patients chronically treated with an antagonist of the renin-angiotensin system. Anesth Analg. 1999 May;88(5):980-4. doi: 10.1097/00000539-199905000-00003. PMID 10320155
- [Background] Giudicelli JF, Berdeaux A, Edouard A, Richer C, Jacolot D. The effect of enalapril on baroreceptor mediated reflex function in normotensive subjects. Br J Clin Pharmacol. 1985 Sep;20(3):211-8. doi: 10.1111/j.1365-2125.1985.tb05063.x. PMID 2994702
- [Background] Gold MI, Abraham EC, Herrington C. A controlled investigation of propofol, thiopentone and methohexitone. Can J Anaesth. 1987 Sep;34(5):478-83. doi: 10.1007/BF03014354. PMID 3499244
- [Background] Komatsu R, You J, Mascha EJ, Sessler DI, Kasuya Y, Turan A. Anesthetic induction with etomidate, rather than propofol, is associated with increased 30-day mortality and cardiovascular morbidity after noncardiac surgery. Anesth Analg. 2013 Dec;117(6):1329-37. doi: 10.1213/ANE.0b013e318299a516. PMID 24257383
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Background] Mets B. Management of hypotension associated with angiotensin-axis blockade and general anesthesia administration. J Cardiothorac Vasc Anesth. 2013 Feb;27(1):156-67. doi: 10.1053/j.jvca.2012.06.014. Epub 2012 Jul 31. No abstract available. PMID 22854335
- [Background] Nielson E, Hennrikus E, Lehman E, Mets B. Angiotensin axis blockade, hypotension, and acute kidney injury in elective major orthopedic surgery. J Hosp Med. 2014 May;9(5):283-8. doi: 10.1002/jhm.2155. Epub 2014 Jan 24. PMID 24464761
- [Background] Price ML, Millar B, Grounds M, Cashman J. Changes in cardiac index and estimated systemic vascular resistance during induction of anaesthesia with thiopentone, methohexitone, propofol and etomidate. Br J Anaesth. 1992 Aug;69(2):172-6. doi: 10.1093/bja/69.2.172. PMID 1389822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 08/2016 through 08/2017 at the pre-anesthesia clinic and on the day of surgery in the pre-operative area.
Period: Overall Study
Arm/Group | Methohexital | Propofol
Started | 26 | 25
Completed | 20 | 25
Not Completed | 6 | 0
Not completed — Physician Decision | 4 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methohexital | Propofol | Total
Number analyzed (Participants) | 20 | 25 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9) | 60 (14) | 61.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 13 | 14 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Hypotensive Events
Description: Hypotensive events under either methohexital or propofol general anesthesia will be counted as the primary outcome measure
Time Frame: Hemodynamic measurements will be taken during the first 15 minutes of anesthetic induction
Measure: Count of Participants; unit: Participants
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 20 | 25
Participants | 8 | 21
Statistical Analysis 1: Comparison: Methohexital vs Propofol; Test type: Superiority; p = 0.01, log-binomial regression — Threshold for significance was p<0.05; Risk Ratio (RR) = 1

2. Secondary Outcome: Number of Participants With Refractory Hypotension
Description: Refractory hypotension is defined as a hypotensive event that continues after 3 doses of vasopressors
Time Frame: Hemodynamic measurements will be taken during the first 15 minutes of anesthetic induction
Measure: Count of Participants; unit: Participants
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 20 | 25
Participants | 2 | 5
Statistical Analysis 1: Comparison: Methohexital vs Propofol; Test type: Superiority; p = 0.37, log binomial regression — Threshold of significance was <0.05; Risk Ratio (RR) = 1

3. Secondary Outcome: Duration of Each Hypotension Episode
Description: This is the length of time that systolic blood pressure was either: (1) < 85 mmHg, or (2) a decrease of more than 30% from the individual's baseline SBP.
Time Frame: Hemodynamic measurements will be taken during the first 15 minutes of anesthetic induction
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 20 | 25
min | 5.1 (3.7) | 4.8 (3.4)

4. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure will be measured through standard monitoring.
Time Frame: Hemodynamic measurements will be taken during the first 15 minutes of anesthetic induction
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 20 | 25
mm Hg | 141 (26) | 126 (22)

5. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure will be measured through standard monitoring.
Time Frame: Hemodynamic measurements will be taken during the first 15 minutes of anesthetic induction
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 20 | 25
mm Hg | 85 (12) | 72 (11)

6. Secondary Outcome: Heart Rate
Description: Heart rate will be measured through standard monitoring.
Time Frame: Hemodynamic measurements will be taken during the first 15 minutes of anesthetic induction
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 20 | 25
bpm | 80 (14) | 76 (15)

7. Secondary Outcome: Serum Concentration of Norepinephrine (NE) (at Baseline (Time 0) and 3,5,10 and 15 Min After Anesthetic Induction)
Description: Serum concentrations of NE at predetermined time points (Baseline (Time 0) and 3,5,10 and 15 min) following anesthetic induction
Time Frame: Time 0,3,5,10 and 15 min following anesthetic induction
Population: Blood samples were not available for some participants at some time points.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 19 | 22
pg/ml
  Time 0: number analyzed (Participants) | 19 | 21
  Time 0 | 205.68 (231.37) | 200.59 (238.26)
  3 min: number analyzed (Participants) | 17 | 22
  3 min | 175.24 (204.52) | 166.04 (222.77)
  5 min: number analyzed (Participants) | 19 | 21
  5 min | 212.34 (230.44) | 208.93 (214.20)
  10 min: number analyzed (Participants) | 19 | 20
  10 min | 179.42 (243.88) | 168.39 (185.79)
  15 min: number analyzed (Participants) | 19 | 20
  15 min | 173.25 (221.62) | 147.32 (163.66)
Statistical Analysis 1: Comparison: Methohexital vs Propofol; Test type: Superiority; p = 0.277, Ratio of Geometric Means — Because the data were skewed, the natural logarithmic transformation was used prior to analysis for inference. Threshold for statistical significance was <0.05; This p-value is for 15 min after induction of anesthesia

8. Secondary Outcome: Blood Levels of Epinephrine (at Baseline (Time 0) and 3,5,10 and 15 Min After Induction of Anesthesia)
Description: Serum concentrations of Epinephrine at predetermined time points (Baseline (Time 0) and 3,5,10 and 15 min) following anesthetic induction
Time Frame: Time 0,3,5,10 and 15 min following anesthetic induction
Population: Blood Samples were not available for some participants at some time points.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 19 | 20
pg/ml
  Time 0: number analyzed (Participants) | 15 | 20
  Time 0 | 70.89 (52.57) | 66.46 (40.82)
  3 min: number analyzed (Participants) | 16 | 20
  3 min | 60.86 (63.46) | 49.87 (34.48)
  5 min | 89.85 (63.52) | 57.29 (31.95)
  10 min: number analyzed (Participants) | 18 | 20
  10 min | 40.96 (36.97) | 44.17 (29.95)
  15 min: number analyzed (Participants) | 15 | 18
  15 min | 46.28 (35.17) | 39.56 (27.77)

9. Secondary Outcome: Blood Levels of Angiotensin II (AII) (at Baseline (Time 0) and 3,5,10 and 15 Min After Anesthetic Induction)
Description: Serum concentrations of Angiotension II at predetermined time points (Baseline (Time 0) and 3,5,10 and 15 min) following anesthetic induction
Time Frame: Time 0,3,5,10 and 15 min following anesthetic induction
Population: Blood samples were not available for some participants at some time points
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 9 | 11
pg/ml
  Time 0 | 21.71 (17.17) | 18.85 (16.15)
  3 min | 19.07 (18.96) | 19.56 (16.84)
  5 min: number analyzed (Participants) | 8 | 10
  5 min | 21.42 (18.70) | 20.62 (15.54)
  10 min: number analyzed (Participants) | 7 | 9
  10 min | 24.46 (17.91) | 20.32 (16.87)
  15 min: number analyzed (Participants) | 6 | 10
  15 min | 22.16 (18.46) | 17.63 (16.42)

10. Secondary Outcome: Blood Levels of Arginine Vasopressin (AVP) (at Baseline (Time 0) and 3,5,10 and 15 Min After Anesthetic Induction) for Participants Who Did Not Receive AVP for Refractory Hypotension
Description: Serum concentrations of AVP at predetermined time points (Baseline (Time 0) and 3,5,10 and 15 min) following anesthetic induction determined for participants who did not receive AVP for refractory hypotension
Time Frame: Time 0,3,5,10 and 15 min following anesthetic induction
Population: Blood samples were not available for some participants at some time points
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 13 | 13
pg/ml
  Time 0: number analyzed (Participants) | 10 | 13
  Time 0 | 30.75 (15.13) | 29.76 (16.17)
  3 min: number analyzed (Participants) | 11 | 12
  3 min | 25.07 (17.41) | 26.50 (16.34)
  5 min: number analyzed (Participants) | 13 | 11
  5 min | 34.66 (19.12) | 23.99 (13.71)
  10 min: number analyzed (Participants) | 12 | 12
  10 min | 29.36 (18.28) | 16.37 (9.18)
  15 min: number analyzed (Participants) | 13 | 10
  15 min | 26.76 (15.00) | 22.15 (7.72)

11. Secondary Outcome: Blood Levels of AVP (at Baseline (Time 0) and 3,5,10 and 15 Min) for Participants Who Received AVP for Refractory Hypotension
Description: Serum concentrations of AVP at predetermined time points (Baseline (Time 0) and 3,5,10 and 15 min), following anesthetic induction, determined for Participants who did not receive AVP for refractory hypotension
Time Frame: Time 0,3,5,10 and 15 min following anesthetic induction
Population: Blood samples were not available for some participants at some time points
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Methohexital | Propofol
Number analyzed (Participants) | 2 | 5
pg/ml
  Time 0 | 14.85 (7.74) | 33.28 (28.96)
  3 min: number analyzed (Participants) | 1 | 5
  3 min | 10.57 | 30.24 (25.13)
  5 min | 13.73 (9.83) | 29.89 (21.28)
  10 min | 13.93 (8.93) | 22.61 (12.25)
  15 min: number analyzed (Participants) | 2 | 3
  15 min | 12.85 (1.22) | 63.86 (45.64)

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Propofol | Methohexital
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT02624050/Prot_SAP_002.pdf
  • Informed Consent Form (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT02624050/ICF_001.pdf